CLINICAL TRIAL: NCT01299480
Title: A Phase 2, Randomized, Placebo-controlled, Single-blind Trial To Assess The Safety, Tolerability, And Immunogenicity Of Bivalent Rlp2086 Vaccine When Administered In Either 2- Or 3-dose Regimens In Healthy Subjects Aged Greater Than Or Equal To 11 To <19 Years
Brief Title: A Trial To Assess The Safety, Tolerability, And Immunogenicity Of Rlp2086 Vaccine When Administered In Either 2- Or 3-Dose Regimens In Healthy Subjects Aged ≥11 To <19 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B1971012; 6108A1-2003 (Other: Alias Study Number); 2009-014493-18 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Meningococcal Vaccine
Keywords: Healthy adolescents
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Experimental): rLP2086 vaccine at visits 1, 2 and 5, saline at visit 3
  Interventions: Biological: Vaccine
- Group 2 (Experimental): rLP2086 vaccine at visits 1, 3, and 5, saline at visit 2
  Interventions: Biological: Vaccine
- Group 3 (Experimental): rLP2086 vaccine at visits 1, and 5, saline at visits 2 and 3
  Interventions: Biological: Vaccine
- Group 4 (Experimental): rLP2086 at visits 1 and 3, saline at visits 2 and 5
  Interventions: Biological: Vaccine
- Group 5 (Experimental): rLP2086 at visits 3 and 5, saline at visits 1 and 2
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — rLP2086 vaccine at visits 1, 2 and 5, saline at visit 3
  Other Names: Group 1
  Arms: Group 1
Biological: Vaccine — rLP2086 vaccine at visits 1, 3, and 5, saline at visit 2
  Other Names: Group 2
  Arms: Group 2
Biological: Vaccine — rLP2086 vaccine at visits 1, and 5, saline at visits 2 and 3
  Other Names: Group 3
  Arms: Group 3
Biological: Vaccine — rLP2086 at visits 1 and 3, saline at visits 2 and 5
  Other Names: Group 4
  Arms: Group 4
Biological: Vaccine — rLP2086 at visits 3 and 5, saline at visits 1 and 2
  Other Names: Group 5
  Arms: Group 5

SUMMARY:
This study is to look at a new vaccine that might prevent meningococcal disease, and to look at the safety of the new vaccine as well as how well it is tolerated. This study will also look at this vaccine being given 2 or 3 times. This study will be done in healthy adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the parent/legally acceptable representative and/or subject has been informed of all pertinent aspects of the study.
* Parent/legally acceptable representative and/or subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Male or female subject aged ≥11 and <19 years at the time of enrollment.
* Available for the entire study period and can be reached by telephone.
* Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
* All male and female subjects must agree to practice a form of effective contraception, such as barrier contraception (ie, condom plus spermicide, a female condom, diaphragm, cervical cap or intrauterine device), implants, injectables, combined oral contraceptives or sexual abstinence prior to entering into the study, for the duration of the vaccination period and for 28 days after the last study vaccination.For Germany: The phrase sexual abstinence is not applicable, with the understanding that all male and all female subjects of childbearing potential must practice an effective form of contraception during the study.
* Negative urine pregnancy test for female subjects.

Exclusion Criteria:

* Previous vaccination with any meningococcal serogroup B vaccine.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* A known or suspected disease of the immune system or those receiving immunosuppressive therapy.
* History of culture-proven disease caused by Neisseria meningitidis or Neisseria gonorrhoeae.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Receipt of any blood products, including immunoglobulin within 6 months before the first study vaccination.
* Current chronic use of systemic antibiotics.
* Participation in other studies during study participation. Participation in purely observational studies is acceptable.
* Received any investigational drugs, vaccines or devices within 28 days before administration of the first study vaccination.
* Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects who are investigational site staff members or subjects who are Pfizer employees directly involved in the conduct of the trial.
* Subject is pregnant or breastfeeding.
* Subject is a direct descendant of study site or Pfizer personnel

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1714 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2012-05-03 (Actual); Study Completion 2012-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- Czechia (13):
  - Ordinace praktickeho lekare pro deti a dorost, Brandýs nad Labem-Stará Boleslav
  - Ordinace praktickeho lekare pro deti a dorost, Chlumec nad Cidlinou
  - Ordinace praktickeho lekare pro deti a dorost, Holice
  - Ordinace praktickeho lekare pro deti a dorost, Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Ordinace praktickeho lekare pro deti a dorost, Odolena Voda
  - Ordinace praktickeho lekare pro deti a dorost, Pardubice
  - Ordinace praktickeho lekare pro deti a dorost, Prague
  - Ordinace praktickeho lekare pro deti a dorost, Praha - Horni Pocernice
  - Ordinace praktickeho lekare pro deti a dorost, Praha - Nusle
  - Ordinace praktickeho lekare pro deti a dorost, Praha 6 - Petriny
  - Ordinace praktickeho lekare pro deti a dorost, Sezemice
- Infektionsmedicinsk Afdeling Q, Aarhus N, Denmark
- Finland (12):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Järvenpää Vaccine Research Clinic, Jarvenpaa
  - Kokkola Vaccine Research Centre, Kokkola
  - Lahti Vaccine Research Clinic, Lahti
  - Oulu Vaccine Research Clinic, Oulu
  - Porin Rokotetutkimusklinikka, Pori
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
  - Vantaa East Vaccine Research Clinic, Vantaa
- Germany (7):
  - Arztpraxis, Bad Saulgau
  - Kinderarzt-Praxis, Bramsche
  - Arztpraxis, Kleve
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Arztpraxis, Neumünster
  - Kinderarztpraxis, Neumünster
  - Kinderarztpraxis, Neustadt/Aisch
- Poland (11):
  - Gabinet Lekarski, Dębica
  - Krakowski Szpital Specjalistyczny, im. Jana Pawla II, Krakow
  - NZOZ "Hipokrates-II" Sp. z o.o., Krakow
  - Nzoz "Anamed" S.C, Lubartów
  - NZOZ Praktyka Lekarza Rodzinnego Eskulap, Lublin
  - NZOZ Praktyka Lekarza Rodzinnego Alina Grocka-Wlazlak, Oborniki Śląskie
  - Specjalistyczny ZOZ nad Matka i Dzieckiem,, Poznan
  - NZLA Michalkowice Jarosz i Partnerzy, Siemianowice Śląskie
  - NZOZ Nasz Lekarz, Torun
  - Szpital im. Sw. Jadwigi Slaskiej, Oddzial Pediatryczny, Trzebnica
  - NZOZ Salmed, Łęczna
- Spain (13):
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Cap Vila Vella, SANT Vicenç DEL Horts, Barcelona
  - Institut Pediatric Mares-Riera, Blanes, Girona
  - Centro de Salud de Paiporta, Paiporta, Valencia
  - Centro de Salud Quart de Poblet, Quart de Poblet, Valencia
  - Hospital Virgen Del Mar, Almería
  - Cap Roquetes-Canteres, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro de Salud Malvarrosa, Valencia
  - Centro Superior de Investigacion en Salud Publica, Valencia
  - Centro Superior de Salud Publica, Valencia
  - Centro de Salud Republica Argentina, Valencia
  - Centro de Salud Trafalgar, Valencia
- Sweden (3):
  - Malarsjukhuset, Infektionsmottagningen, Eskilstuna
  - Skanes Universitetssjukhus Malmo, Barn- och Ungdomscentrum, Malmo
  - CRS, Clinical Research Support, Örebro

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Beeslaar J, Peyrani P, Absalon J, Maguire J, Eiden J, Balmer P, Maansson R, Perez JL. Sex, Age, and Race Effects on Immunogenicity of MenB-FHbp, A Bivalent Meningococcal B Vaccine: Pooled Evaluation of Clinical Trial Data. Infect Dis Ther. 2020 Sep;9(3):625-639. doi: 10.1007/s40121-020-00322-5. Epub 2020 Jul 17. PMID 32681472
- [Derived] Vesikari T, Ostergaard L, Diez-Domingo J, Wysocki J, Flodmark CE, Beeslaar J, Eiden J, Jiang Q, Jansen KU, Jones TR, Harris SL, O'Neill RE, York LJ, Crowther G, Perez JL. Meningococcal Serogroup B Bivalent rLP2086 Vaccine Elicits Broad and Robust Serum Bactericidal Responses in Healthy Adolescents. J Pediatric Infect Dis Soc. 2016 Jun;5(2):152-60. doi: 10.1093/jpids/piv039. Epub 2015 Aug 4. PMID 26407272

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1714 participants were enrolled in this study. Of these, 1 participant was not randomized but was vaccinated with Saline at Injection 1. This participant was included in safety population and not intent-to-treat population. Participant Flow includes only randomized intent to treat participants.
Groups:
- Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month): Randomized to receive rLP2086 on a 0-, 1-, 6- month and 0.9% normal saline on a 2- month schedule.
- Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month): Randomized to receive rLP2086 on a 0-, 2-, 6- month and 0.9% normal saline on a 1- month schedule.
- Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month): Randomized to receive rLP2086 on a 0-, 6- month and 0.9% normal saline on a 1-, 2- month schedule.
- Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month): Randomized to receive rLP2086 on a 0-, 2- month and 0.9% normal saline on a 1-, 6- month schedule.
- Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month): Randomized to receive rLP2086 on a 2-, 6- month and 0.9% normal saline on a 0-, 1- month schedule.
Period: Overall Study
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month)
Started | 427 | 430 | 427 | 286 | 143
Completed | 385 | 395 | 386 | 261 | 123
Not Completed | 42 | 35 | 41 | 25 | 20
Not completed — No longer willing to participate | 19 | 17 | 14 | 13 | 10
Not completed — Protocol Violation | 7 | 5 | 8 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 4 | 7 | 3 | 4
Not completed — Adverse Event | 6 | 4 | 5 | 4 | 0
Not completed — Withdrawal due to pregnancy | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 3 | 1 | 2 | 1 | 2
Not completed — Other | 3 | 2 | 3 | 0 | 3
Not completed — Started, but not vaccinated | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month) | Total
Number analyzed (Participants) | 427 | 430 | 427 | 286 | 143 | 1713
Age, Customized [Number; unit: participants]
  11- less than (<) 14 years | 156 | 158 | 156 | 106 | 53 | 629
  14 - <19 years | 271 | 272 | 271 | 180 | 90 | 1084
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 225 | 216 | 139 | 79 | 871
  Male | 215 | 205 | 211 | 147 | 64 | 842

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serum Bactericidal Assay Using Human Complement (hSBA) Titer Greater Than or Equal to (>=) Lower Limit of Quantitation: Group 1 and 2 Participants
Time Frame: 1 month after Injection 4
Population: The number of participants shown for each test strain represents the number with valid and determinant assay result for that strain.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month)
Number analyzed (Participants) | 365 | 360
percentage of participants
  PMB80 [A22] 1:8 (N=360, 357): number analyzed (Participants) | 360 | 357
  PMB80 [A22] 1:8 (N=360, 357) | 91.7 | 95.0
  PMB2001 [A56] 1:8 (N=362, 359): number analyzed (Participants) | 362 | 359
  PMB2001 [A56] 1:8 (N=362, 359) | 99.4 | 98.9
  PMB2948 [B24] 1:8 (N=354, 354): number analyzed (Participants) | 354 | 354
  PMB2948 [B24] 1:8 (N=354, 354) | 89.0 | 88.4
  PMB2707 [B44] 1:8 (N356, 352): number analyzed (Participants) | 356 | 352
  PMB2707 [B44] 1:8 (N356, 352) | 88.5 | 86.1
Statistical Analysis 1: Comparison: Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month); PMB80 [A22]: Response rate was compared with 50%, using 1-sided exact test based on binomial distribution. p-Value <0.0125 was considered significant; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 2: Comparison: Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month); PMB2001 [A56]: Response rate was compared with 50%, using 1-sided exact test based on binomial distribution. p-Value <0.0125 was considered significant; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 3: Comparison: Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month); PMB2948 [B24]: Response rate was compared with 50%, using 1-sided exact test based on binomial distribution. p-Value <0.0125 was considered significant; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 4: Comparison: Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month); PMB2707 [B44]: Response rate was compared with 50%, using 1-sided exact test based on binomial distribution. p-Value <0.0125 was considered significant; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 5: Comparison: Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 6: Comparison: Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 7: Comparison: Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 8: Comparison: Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.001, Binomial Distribution

2. Primary Outcome: Percentage of Participants Reporting At Least 1 Adverse Event (AE)
Time Frame: Injection 1 up to 1 month after Injection 4
Population: Some participants randomized to receive vaccination as per Groups 1, 2 or 4 schedules actually received vaccination as per Group 3 schedule. One participant was not randomized but received Saline at Injection 1 and was included in Group 5. Participants have been presented as per actual administration schedule received.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month)
Number analyzed (Participants) | 426 | 414 | 451 | 277 | 144
percentage of participants | 36.9 | 35.7 | 35.5 | 35.7 | 37.5

3. Secondary Outcome: Percentage of Participants Achieving hSBA Titer >=LLOQ: Group 3 Participants
Time Frame: 1 month after Injection 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month)
Number analyzed (Participants) | 371
percentage of participants
  PMB80 [A22] 1:8 (N=369): number analyzed (Participants) | 369
  PMB80 [A22] 1:8 (N=369) | 93.5
  PMB2001 [A56] 1: 8 (N=370): number analyzed (Participants) | 370
  PMB2001 [A56] 1: 8 (N=370) | 98.4
  PMB2948 [B24] 1:8 (N=359): number analyzed (Participants) | 359
  PMB2948 [B24] 1:8 (N=359) | 81.1
  PMB2707 [B44] 1:8 (N=356): number analyzed (Participants) | 356
  PMB2707 [B44] 1:8 (N=356) | 77.5
Statistical Analysis 1: Comparison: Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 2: Comparison: Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 3: Comparison: Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Binomial Distribution
Statistical Analysis 4: Comparison: Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.001, Binomial Distribution

4. Secondary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) Geometric Mean Titers (GMTs)
Time Frame: Before Injection (Inj) 1, 1 Month (M) after (aft) Injection 2, 3, 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month)
Number analyzed (Participants) | 365 | 360 | 371 | 241 | 113
titer
  Before Inj1: PMB80 [A22]; N=356,352,364,235,108: number analyzed (Participants) | 356 | 352 | 364 | 235 | 108
  Before Inj1: PMB80 [A22]; N=356,352,364,235,108 | 7.1 [6.41 to 7.87] | 6.3 [5.72 to 6.95] | 6.4 [5.84 to 7.02] | 6.4 [5.66 to 7.22] | 6.8 [5.59 to 8.30]
  1M aft Inj2: PMB80 [A22]; N=351,345,351,224,110: number analyzed (Participants) | 351 | 345 | 351 | 224 | 110
  1M aft Inj2: PMB80 [A22]; N=351,345,351,224,110 | 24.4 [21.25 to 27.94] | 10.7 [9.44 to 12.09] | 12.0 [10.58 to 13.60] | 13.3 [11.21 to 15.76] | 7.1 [5.86 to 8.48]
  1M aft Inj3: PMB80 [A22]; N=332,344,340,238,102: number analyzed (Participants) | 332 | 344 | 340 | 238 | 102
  1M aft Inj3: PMB80 [A22]; N=332,344,340,238,102 | 17.7 [15.28 to 20.47] | 32.9 [29.34 to 36.92] | 10.3 [9.09 to 11.68] | 37.1 [32.23 to 42.76] | 16.0 [12.15 to 21.06]
  1M aft Inj4: PMB80 [A22]; N=360,357,369,234,111: number analyzed (Participants) | 360 | 357 | 369 | 234 | 111
  1M aft Inj4: PMB80 [A22]; N=360,357,369,234,111 | 55.1 [48.87 to 62.07] | 56.3 [50.91 to 62.27] | 48.4 [43.45 to 53.86] | 14.2 [12.08 to 16.73] | 39.6 [32.31 to 48.46]
  Before Inj1: PMB2001 [A56]; N=350,348,355,231,107: number analyzed (Participants) | 350 | 348 | 355 | 231 | 107
  Before Inj1: PMB2001 [A56]; N=350,348,355,231,107 | 6.8 [6.06 to 7.64] | 6.1 [5.54 to 6.77] | 6.7 [6.00 to 7.48] | 6.3 [5.54 to 7.15] | 6.2 [5.10 to 7.47]
  1M aft Inj2: PMB2001 [A56]; N=353,329,335,218,102: number analyzed (Participants) | 353 | 329 | 335 | 218 | 102
  1M aft Inj2: PMB2001 [A56]; N=353,329,335,218,102 | 77.3 [68.54 to 87.12] | 17.0 [14.56 to 19.96] | 18.5 [15.81 to 21.63] | 17.7 [14.45 to 21.58] | 6.8 [5.52 to 8.36]
  1M aft Inj3: PMB2001 [A56]; N=329,339,320,240,102: number analyzed (Participants) | 329 | 339 | 320 | 240 | 102
  1M aft Inj3: PMB2001 [A56]; N=329,339,320,240,102 | 48.3 [41.96 to 55.50] | 94.6 [84.64 to 105.68] | 15.1 [12.89 to 17.74] | 104.9 [93.16 to 118.05] | 26.8 [19.48 to 36.92]
  1M aft Inj4: PMB2001 [A56]; N=362,359,370,228,113: number analyzed (Participants) | 362 | 359 | 370 | 228 | 113
  1M aft Inj4: PMB2001 [A56]; N=362,359,370,228,113 | 152.9 [137.23 to 170.47] | 155.6 [140.39 to 172.38] | 125.6 [112.59 to 140.17] | 26.5 [22.24 to 31.58] | 111.8 [92.73 to 134.90]
  Before Inj1: PMB2948 [B24]; N=362,356,369,241,112: number analyzed (Participants) | 362 | 356 | 369 | 241 | 112
  Before Inj1: PMB2948 [B24]; N=362,356,369,241,112 | 5.3 [4.93 to 5.75] | 5.1 [4.77 to 5.52] | 5.0 [4.70 to 5.38] | 4.9 [4.49 to 5.24] | 5.1 [4.51 to 5.82]
  1M aft Inj2: PMB2948 [B24]; N=344,345,352,223,110: number analyzed (Participants) | 344 | 345 | 352 | 223 | 110
  1M aft Inj2: PMB2948 [B24]; N=344,345,352,223,110 | 13.8 [12.15 to 15.57] | 8.2 [7.38 to 9.21] | 9.2 [8.20 to 10.28] | 9.8 [8.39 to 11.35] | 5.3 [4.70 to 6.08]
  1M aft Inj3: PMB2948 [B24]; N=328,337,340,237,102: number analyzed (Participants) | 328 | 337 | 340 | 237 | 102
  1M aft Inj3: PMB2948 [B24]; N=328,337,340,237,102 | 11.0 [9.61 to 12.50] | 14.9 [13.20 to 16.73] | 7.5 [6.75 to 8.35] | 17.7 [15.24 to 20.49] | 12.6 [10.01 to 15.89]
  1M aft Inj4: PMB2948 [B24]; N=354,354,359,228,110: number analyzed (Participants) | 354 | 354 | 359 | 228 | 110
  1M aft Inj4: PMB2948 [B24]; N=354,354,359,228,110 | 29.1 [25.88 to 32.66] | 25.6 [23.03 to 28.45] | 20.6 [18.38 to 23.18] | 8.0 [7.01 to 9.24] | 14.7 [12.01 to 18.10]
  Before Inj1: PMB2707 [B44]; N=363,357,370,241,113: number analyzed (Participants) | 363 | 357 | 370 | 241 | 113
  Before Inj1: PMB2707 [B44]; N=363,357,370,241,113 | 4.4 [4.18 to 4.54] | 4.5 [4.24 to 4.67] | 4.5 [4.26 to 4.70] | 4.6 [4.28 to 4.90] | 4.4 [4.04 to 4.76]
  1M aft Inj2: PMB2707 [B44]; N=341,345,349,225,111: number analyzed (Participants) | 341 | 345 | 349 | 225 | 111
  1M aft Inj2: PMB2707 [B44]; N=341,345,349,225,111 | 13.1 [11.29 to 15.11] | 5.5 [5.04 to 6.01] | 5.7 [5.19 to 6.30] | 5.9 [5.19 to 6.74] | 4.4 [4.04 to 4.77]
  1M aft Inj3: PMB2707 [B44]; N=333,331,341,234,105: number analyzed (Participants) | 333 | 331 | 341 | 234 | 105
  1M aft Inj3: PMB2707 [B44]; N=333,331,341,234,105 | 8.4 [7.40 to 9.60] | 15.5 [13.51 to 17.87] | 5.2 [4.78 to 5.68] | 19.1 [16.03 to 22.78] | 6.8 [5.45 to 8.55]
  1M aft Inj4: PMB2707 [B44]; N=356,352,356,230,111: number analyzed (Participants) | 356 | 352 | 356 | 230 | 111
  1M aft Inj4: PMB2707 [B44]; N=356,352,356,230,111 | 40.3 [35.16 to 46.11] | 35.0 [30.63 to 39.91] | 22.5 [19.60 to 25.72] | 6.2 [5.52 to 7.07] | 17.8 [14.12 to 22.42]

5. Secondary Outcome: Percentage of Participants Achieving hSBA Titer >=LLOQ
Time Frame: Before Injection 1, 1 Month after Injection 2, 3, 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month)
Number analyzed (Participants) | 365 | 360 | 371 | 241 | 113
percentage of participants
  Before Inj1: PMB80[A22] 1:8; N=356,352,364,235,108: number analyzed (Participants) | 356 | 352 | 364 | 235 | 108
  Before Inj1: PMB80[A22] 1:8; N=356,352,364,235,108 | 28.1 | 21.9 | 24.7 | 22.6 | 25.0
  1M aft Inj2:PMB80[A22]1:8; N=351,345,351,224,110: number analyzed (Participants) | 351 | 345 | 351 | 224 | 110
  1M aft Inj2:PMB80[A22]1:8; N=351,345,351,224,110 | 74.6 | 46.7 | 51.3 | 52.2 | 28.2
  1M aft Inj3:PMB80[A22]1:8; N=332,344,340,238,102: number analyzed (Participants) | 332 | 344 | 340 | 238 | 102
  1M aft Inj3:PMB80[A22]1:8; N=332,344,340,238,102 | 63.0 | 88.7 | 44.7 | 90.8 | 55.9
  1M aft Inj4:PMB80[A22]1:8; N=360,357,369,234,111: number analyzed (Participants) | 360 | 357 | 369 | 234 | 111
  1M aft Inj4:PMB80[A22]1:8; N=360,357,369,234,111 | 91.7 | 95.0 | 93.5 | 57.7 | 91.9
  Before Inj1:PMB2001[A56]1:8; N=350,348,355,231,107: number analyzed (Participants) | 350 | 348 | 355 | 231 | 107
  Before Inj1:PMB2001[A56]1:8; N=350,348,355,231,107 | 20.9 | 18.7 | 21.7 | 19.0 | 17.8
  1M aft Inj2:PMB2001[A56]1:8; N=353,329,335,218,102: number analyzed (Participants) | 353 | 329 | 335 | 218 | 102
  1M aft Inj2:PMB2001[A56]1:8; N=353,329,335,218,102 | 96.6 | 56.2 | 58.8 | 56.0 | 22.5
  1M aft Inj3;PMB2001[A56]1:8; N=329,339,320,240,102: number analyzed (Participants) | 329 | 339 | 320 | 240 | 102
  1M aft Inj3;PMB2001[A56]1:8; N=329,339,320,240,102 | 89.1 | 97.9 | 50.6 | 100.0 | 67.6
  1M aft Inj4:PMB2001[A56]1:8; N=362,359,370,228,113: number analyzed (Participants) | 362 | 359 | 370 | 228 | 113
  1M aft Inj4:PMB2001[A56]1:8; N=362,359,370,228,113 | 99.4 | 98.9 | 98.4 | 76.8 | 99.1
  Before Inj1:PMB2948[B24]1:8; N=362,356,369,241,112: number analyzed (Participants) | 362 | 356 | 369 | 241 | 112
  Before Inj1:PMB2948[B24]1:8; N=362,356,369,241,112 | 16.3 | 13.8 | 13.0 | 11.2 | 14.3
  1M aft Inj2:PMB2948[B24]1:8; N=344,345,352,223,110: number analyzed (Participants) | 344 | 345 | 352 | 223 | 110
  1M aft Inj2:PMB2948[B24]1:8; N=344,345,352,223,110 | 62.2 | 39.4 | 43.8 | 45.3 | 18.2
  1M aft Inj3:PMB2948[B24]1:8; N=328,337,340,237,102: number analyzed (Participants) | 328 | 337 | 340 | 237 | 102
  1M aft Inj3:PMB2948[B24]1:8; N=328,337,340,237,102 | 50.6 | 70.3 | 35.6 | 73.0 | 56.9
  1M aft Inj4:PMB2948[B24]1:8; N=354,354,359,228,110: number analyzed (Participants) | 354 | 354 | 359 | 228 | 110
  1M aft Inj4:PMB2948[B24]1:8; N=354,354,359,228,110 | 89.0 | 88.4 | 81.1 | 35.5 | 69.1
  Before Inj1:PMB2707[B44]1:8; N=363,357,370,241,113: number analyzed (Participants) | 363 | 357 | 370 | 241 | 113
  Before Inj1:PMB2707[B44]1:8; N=363,357,370,241,113 | 5.2 | 6.2 | 6.2 | 7.5 | 4.4
  1M aft Inj2:PMB2707[B44]1:8; N=341,345,349,225,111: number analyzed (Participants) | 341 | 345 | 349 | 225 | 111
  1M aft Inj2:PMB2707[B44]1:8; N=341,345,349,225,111 | 54.0 | 15.7 | 17.8 | 18.2 | 4.5
  1M aft Inj3:PMB2707[B44]1:8; N=333,331,341,234,105: number analyzed (Participants) | 333 | 331 | 341 | 234 | 105
  1M aft Inj3:PMB2707[B44]1:8; N=333,331,341,234,105 | 35.4 | 61.9 | 12.6 | 70.1 | 23.8
  1M aft Inj4:PMB2707[B44]1:8; N=356,352,356,230,111: number analyzed (Participants) | 356 | 352 | 356 | 230 | 111
  1M aft Inj4:PMB2707[B44]1:8; N=356,352,356,230,111 | 88.5 | 86.1 | 77.5 | 23.9 | 73.0

6. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer >= Prespecified Titer Level
Time Frame: Before Injection 1, 1 Month after Injection 2, 3, 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month)
Number analyzed (Participants) | 365 | 360 | 371 | 241 | 113
percentage of participants
  Before Inj1:PMB80[A22] 1:4; N=356,352,364,235,108: number analyzed (Participants) | 356 | 352 | 364 | 235 | 108
  Before Inj1:PMB80[A22] 1:4; N=356,352,364,235,108 | 28.9 | 23.9 | 26.4 | 23.8 | 25.9
  Before Inj1:PMB80[A22] 1:16; N=356,352,364,235,108: number analyzed (Participants) | 356 | 352 | 364 | 235 | 108
  Before Inj1:PMB80[A22] 1:16; N=356,352,364,235,108 | 27.2 | 20.5 | 22.8 | 22.1 | 24.1
  Before Inj1:PMB80[A22] 1:32; N=356,352,364,235,108: number analyzed (Participants) | 356 | 352 | 364 | 235 | 108
  Before Inj1:PMB80[A22] 1:32; N=356,352,364,235,108 | 18.3 | 14.5 | 13.5 | 13.2 | 15.7
  Before Inj1:PMB80[A22] 1:64; N=356,352,364,235,108: number analyzed (Participants) | 356 | 352 | 364 | 235 | 108
  Before Inj1:PMB80[A22] 1:64; N=356,352,364,235,108 | 7.6 | 6.5 | 4.7 | 6.8 | 7.4
  Before Inj1:PMB80[A22]1:128; N=356,352,364,235,108: number analyzed (Participants) | 356 | 352 | 364 | 235 | 108
  Before Inj1:PMB80[A22]1:128; N=356,352,364,235,108 | 1.4 | 2.3 | 1.6 | 2.6 | 1.9
  1M aft Inj2:PMB80[A22] 1:4; N=351,345,351,224,110: number analyzed (Participants) | 351 | 345 | 351 | 224 | 110
  1M aft Inj2:PMB80[A22] 1:4; N=351,345,351,224,110 | 74.9 | 47.8 | 51.3 | 52.2 | 29.1
  1M aft Inj2:PMB80[A22] 1:16; N=351,345,351,224,110: number analyzed (Participants) | 351 | 345 | 351 | 224 | 110
  1M aft Inj2:PMB80[A22] 1:16; N=351,345,351,224,110 | 73.5 | 45.8 | 50.7 | 51.8 | 27.3
  1M aft Inj2:PMB80[A22] 1:32; N=351,345,351,224,110: number analyzed (Participants) | 351 | 345 | 351 | 224 | 110
  1M aft Inj2:PMB80[A22] 1:32; N=351,345,351,224,110 | 58.4 | 28.7 | 34.5 | 37.9 | 18.2
  1M aft Inj2:PMB80[A22] 1:64; N=351,345,351,224,110: number analyzed (Participants) | 351 | 345 | 351 | 224 | 110
  1M aft Inj2:PMB80[A22] 1:64; N=351,345,351,224,110 | 30.8 | 14.5 | 14.5 | 19.6 | 6.4
  1M aft Inj2:PMB80[A22]1:128; N=351,345,351,224,110: number analyzed (Participants) | 351 | 345 | 351 | 224 | 110
  1M aft Inj2:PMB80[A22]1:128; N=351,345,351,224,110 | 14.8 | 5.2 | 5.7 | 8.5 | 0.9
  1M aft Inj3:PMB80[A22] 1:4; N=332,344,340,238,102: number analyzed (Participants) | 332 | 344 | 340 | 238 | 102
  1M aft Inj3:PMB80[A22] 1:4; N=332,344,340,238,102 | 63.6 | 88.7 | 45.6 | 90.8 | 55.9
  1M aft Inj3:PMB80[A22]1:16; N=332,344,340,238,102: number analyzed (Participants) | 332 | 344 | 340 | 238 | 102
  1M aft Inj3:PMB80[A22]1:16; N=332,344,340,238,102 | 62.3 | 88.1 | 42.4 | 90.8 | 55.9
  1M aft Inj3:PMB80[A22]1:32; N=332,344,340,238,102: number analyzed (Participants) | 332 | 344 | 340 | 238 | 102
  1M aft Inj3:PMB80[A22]1:32; N=332,344,340,238,102 | 47.3 | 69.5 | 30.6 | 70.6 | 45.1
  1M aft Inj3:PMB80[A22]1:64; N=332,344,340,238,102: number analyzed (Participants) | 332 | 344 | 340 | 238 | 102
  1M aft Inj3:PMB80[A22]1:64; N=332,344,340,238,102 | 22.3 | 35.8 | 12.4 | 39.1 | 22.5
  1M aft Inj3:PMB80[A22]1:128; N=332,344,340,238,102: number analyzed (Participants) | 332 | 344 | 340 | 238 | 102
  1M aft Inj3:PMB80[A22]1:128; N=332,344,340,238,102 | 11.7 | 14.8 | 4.4 | 19.7 | 14.7
  1M aft Inj4:PMB80[A22] 1:4; N=360,357,369,234,111: number analyzed (Participants) | 360 | 357 | 369 | 234 | 111
  1M aft Inj4:PMB80[A22] 1:4; N=360,357,369,234,111 | 91.9 | 95.0 | 94.0 | 58.1 | 91.9
  1M aft Inj4:PMB80[A22] 1:16; N=360,357,369,234,111: number analyzed (Participants) | 360 | 357 | 369 | 234 | 111
  1M aft Inj4:PMB80[A22] 1:16; N=360,357,369,234,111 | 91.4 | 95.0 | 93.2 | 56.0 | 91.0
  1M aft Inj4:PMB80[A22] 1:32; N=360,357,369,234,111: number analyzed (Participants) | 360 | 357 | 369 | 234 | 111
  1M aft Inj4:PMB80[A22] 1:32; N=360,357,369,234,111 | 84.2 | 86.6 | 81.8 | 38.0 | 74.8
  1M aft Inj4:PMB80[A22] 1:64; N=360,357,369,234,111: number analyzed (Participants) | 360 | 357 | 369 | 234 | 111
  1M aft Inj4:PMB80[A22] 1:64; N=360,357,369,234,111 | 61.9 | 63.9 | 53.9 | 19.2 | 42.3
  1M aft Inj4:PMB80[A22]1:128; N=360,357,369,234,111: number analyzed (Participants) | 360 | 357 | 369 | 234 | 111
  1M aft Inj4:PMB80[A22]1:128; N=360,357,369,234,111 | 31.7 | 32.5 | 25.7 | 8.5 | 20.7
  Before Inj1:PMB2001[A56] 1:4;N=350,348,355,231,107: number analyzed (Participants) | 350 | 348 | 355 | 231 | 107
  Before Inj1:PMB2001[A56] 1:4;N=350,348,355,231,107 | 25.1 | 22.1 | 25.1 | 25.5 | 25.2
  Before Inj1:PMB2001[A56]1:16;N=350,348,355,231,107: number analyzed (Participants) | 350 | 348 | 355 | 231 | 107
  Before Inj1:PMB2001[A56]1:16;N=350,348,355,231,107 | 20.0 | 18.1 | 20.3 | 19.0 | 16.8
  Before Inj1:PMB2001[A56]1:32;N=350,348,355,231,107: number analyzed (Participants) | 350 | 348 | 355 | 231 | 107
  Before Inj1:PMB2001[A56]1:32;N=350,348,355,231,107 | 18.0 | 14.1 | 17.2 | 15.6 | 15.9
  Before Inj1:PMB2001[A56]1:64;N=350,348,355,231,107: number analyzed (Participants) | 350 | 348 | 355 | 231 | 107
  Before Inj1:PMB2001[A56]1:64;N=350,348,355,231,107 | 11.7 | 7.5 | 10.7 | 8.7 | 8.4
  Before Inj1: PMB2001 1:128;N=350,348,355,231,107: number analyzed (Participants) | 350 | 348 | 355 | 231 | 107
  Before Inj1: PMB2001 1:128;N=350,348,355,231,107 | 4.3 | 2.3 | 3.7 | 2.6 | 2.8
  1M aft Inj2:PMB2001[A56] 1:4;N=353,329,335,218,102: number analyzed (Participants) | 353 | 329 | 335 | 218 | 102
  1M aft Inj2:PMB2001[A56] 1:4;N=353,329,335,218,102 | 96.6 | 61.4 | 63.3 | 60.1 | 25.5
  1M aft Inj2:PMB2001[A56]1:16;N=353,329,335,218,102: number analyzed (Participants) | 353 | 329 | 335 | 218 | 102
  1M aft Inj2:PMB2001[A56]1:16;N=353,329,335,218,102 | 96.3 | 55.0 | 57.9 | 55.5 | 21.6
  1M aft Inj2:PMB2001[A56]1:32;N=353,329,335,218,102: number analyzed (Participants) | 353 | 329 | 335 | 218 | 102
  1M aft Inj2:PMB2001[A56]1:32;N=353,329,335,218,102 | 87.8 | 48.0 | 50.1 | 47.2 | 17.6
  1M aft Inj2:PMB2001[A56]1:64;N=353,329,335,218,102: number analyzed (Participants) | 353 | 329 | 335 | 218 | 102
  1M aft Inj2:PMB2001[A56]1:64;N=353,329,335,218,102 | 72.8 | 27.4 | 31.0 | 29.8 | 10.8
  1M aft Inj2:PMB2001 1:128;N=353,329,335,218,102: number analyzed (Participants) | 353 | 329 | 335 | 218 | 102
  1M aft Inj2:PMB2001 1:128;N=353,329,335,218,102 | 41.1 | 14.3 | 14.9 | 15.6 | 2.9
  1M aft Inj3:PMB2001[A56] 1:4;N=329,339,320,240,102: number analyzed (Participants) | 329 | 339 | 320 | 240 | 102
  1M aft Inj3:PMB2001[A56] 1:4;N=329,339,320,240,102 | 91.5 | 98.5 | 54.4 | 100.0 | 72.5
  1M aft Inj3:PMB2001[A56]1:16;N=329,339,320,240,102: number analyzed (Participants) | 329 | 339 | 320 | 240 | 102
  1M aft Inj3:PMB2001[A56]1:16;N=329,339,320,240,102 | 87.8 | 97.9 | 50.0 | 99.2 | 65.7
  1M aft Inj3:PMB2001[A56]1:32;N=329,339,320,240,102: number analyzed (Participants) | 329 | 339 | 320 | 240 | 102
  1M aft Inj3:PMB2001[A56]1:32;N=329,339,320,240,102 | 79.9 | 94.1 | 43.8 | 95.0 | 55.9
  1M aft Inj3:PMB2001[A56]1:64;N=329,339,320,240,102: number analyzed (Participants) | 329 | 339 | 320 | 240 | 102
  1M aft Inj3:PMB2001[A56]1:64;N=329,339,320,240,102 | 52.9 | 79.1 | 28.4 | 81.7 | 39.2
  1M aft Inj3:PMB2001 1:128;N=329,339,320,240,102: number analyzed (Participants) | 329 | 339 | 320 | 240 | 102
  1M aft Inj3:PMB2001 1:128;N=329,339,320,240,102 | 26.7 | 50.4 | 13.1 | 57.1 | 22.5
  1M aft Inj4:PMB2001[A56] 1:4;N=362,359,370,228,113: number analyzed (Participants) | 362 | 359 | 370 | 228 | 113
  1M aft Inj4:PMB2001[A56] 1:4;N=362,359,370,228,113 | 99.7 | 99.2 | 98.9 | 79.8 | 99.1
  1M aft Inj4:PMB2001[A56]1:16;N=362,359,370,228,113: number analyzed (Participants) | 362 | 359 | 370 | 228 | 113
  1M aft Inj4:PMB2001[A56]1:16;N=362,359,370,228,113 | 99.2 | 98.9 | 98.4 | 74.6 | 99.1
  1M aft Inj4:PMB2001[A56]1:32;N=362,359,370,228,113: number analyzed (Participants) | 362 | 359 | 370 | 228 | 113
  1M aft Inj4:PMB2001[A56]1:32;N=362,359,370,228,113 | 95.3 | 96.1 | 94.6 | 59.6 | 92.9
  1M aft Inj4:PMB2001[A56]1:64;N=362,359,370,228,113: number analyzed (Participants) | 362 | 359 | 370 | 228 | 113
  1M aft Inj4:PMB2001[A56]1:64;N=362,359,370,228,113 | 87.8 | 91.1 | 83.8 | 34.2 | 85.0
  1M aft Inj4:PMB2001 1:128;N=362,359,370,228,113: number analyzed (Participants) | 362 | 359 | 370 | 228 | 113
  1M aft Inj4:PMB2001 1:128;N=362,359,370,228,113 | 72.4 | 73.5 | 65.9 | 15.8 | 60.2
  Before Inj1:PMB2948[B24]1:4;N=362,356,369,241,112: number analyzed (Participants) | 362 | 356 | 369 | 241 | 112
  Before Inj1:PMB2948[B24]1:4;N=362,356,369,241,112 | 18.5 | 15.4 | 14.4 | 13.3 | 16.1
  Before Inj1:PMB2948[B24]1:16;N=362,356,369,241,112: number analyzed (Participants) | 362 | 356 | 369 | 241 | 112
  Before Inj1:PMB2948[B24]1:16;N=362,356,369,241,112 | 12.7 | 11.5 | 10.8 | 8.7 | 12.5
  Before Inj1:PMB2948[B24]1:32;N=362,356,369,241,112: number analyzed (Participants) | 362 | 356 | 369 | 241 | 112
  Before Inj1:PMB2948[B24]1:32;N=362,356,369,241,112 | 7.2 | 6.2 | 6.0 | 5.0 | 4.5
  Before Inj1:PMB2948[B24]1:64;N=362,356,369,241,112: number analyzed (Participants) | 362 | 356 | 369 | 241 | 112
  Before Inj1:PMB2948[B24]1:64;N=362,356,369,241,112 | 2.8 | 3.1 | 2.2 | 2.1 | 2.7
  Before Inj1:PMB2948 1:128;N=362,356,369,241,112: number analyzed (Participants) | 362 | 356 | 369 | 241 | 112
  Before Inj1:PMB2948 1:128;N=362,356,369,241,112 | 1.4 | 0.8 | 0.5 | 0.8 | 1.8
  1M aft Inj2:PMB2948[B24]1:4;N=344,345,352,223,110: number analyzed (Participants) | 344 | 345 | 352 | 223 | 110
  1M aft Inj2:PMB2948[B24]1:4;N=344,345,352,223,110 | 66.3 | 42.3 | 45.7 | 47.1 | 20.0
  1M aft Inj2:PMB2948[B24]1:16;N=344,345,352,223,110: number analyzed (Participants) | 344 | 345 | 352 | 223 | 110
  1M aft Inj2:PMB2948[B24]1:16;N=344,345,352,223,110 | 57.6 | 32.8 | 39.5 | 40.4 | 14.5
  1M aft Inj2:PMB2948[B24]1:32;N=344,345,352,223,110: number analyzed (Participants) | 344 | 345 | 352 | 223 | 110
  1M aft Inj2:PMB2948[B24]1:32;N=344,345,352,223,110 | 34.9 | 18.6 | 23.3 | 24.7 | 5.5
  1M aft Inj2:PMB2948[B24]1:64;N=344,345,352,223,110: number analyzed (Participants) | 344 | 345 | 352 | 223 | 110
  1M aft Inj2:PMB2948[B24]1:64;N=344,345,352,223,110 | 14.0 | 9.0 | 8.8 | 11.7 | 3.6
  1M aft Inj2:PMB2948 1:128;N=344,345,352,223,110: number analyzed (Participants) | 344 | 345 | 352 | 223 | 110
  1M aft Inj2:PMB2948 1:128;N=344,345,352,223,110 | 6.1 | 3.5 | 2.6 | 4.5 | 0.0
  1M aft Inj3:PMB2948[B24]1:4;N=328,337,340,237,102: number analyzed (Participants) | 328 | 337 | 340 | 237 | 102
  1M aft Inj3:PMB2948[B24]1:4;N=328,337,340,237,102 | 52.1 | 72.1 | 37.6 | 75.5 | 57.8
  1M aft Inj3:PMB2948[B24]1:16;N=328,337,340,237,102: number analyzed (Participants) | 328 | 337 | 340 | 237 | 102
  1M aft Inj3:PMB2948[B24]1:16;N=328,337,340,237,102 | 45.1 | 63.5 | 29.7 | 67.1 | 52.9
  1M aft Inj3:PMB2948[B24]1:32;N=328,337,340,237,102: number analyzed (Participants) | 328 | 337 | 340 | 237 | 102
  1M aft Inj3:PMB2948[B24]1:32;N=328,337,340,237,102 | 23.8 | 32.0 | 15.9 | 43.5 | 32.4
  1M aft Inj3:PMB2948[B24]1:64;N=328,337,340,237,102: number analyzed (Participants) | 328 | 337 | 340 | 237 | 102
  1M aft Inj3:PMB2948[B24]1:64;N=328,337,340,237,102 | 15.5 | 13.6 | 5.0 | 19.4 | 15.7
  1M aft Inj3:PMB2948 1:128;N=328,337,340,237,102: number analyzed (Participants) | 328 | 337 | 340 | 237 | 102
  1M aft Inj3:PMB2948 1:128;N=328,337,340,237,102 | 6.7 | 6.5 | 2.6 | 8.4 | 6.9
  1M aft Inj4:PMB2948[B24]1:4;N=354,354,359,228,110: number analyzed (Participants) | 354 | 354 | 359 | 228 | 110
  1M aft Inj4:PMB2948[B24]1:4;N=354,354,359,228,110 | 90.1 | 90.1 | 83.0 | 38.2 | 70.9
  1M aft Inj4:PMB2948[B24]1:16;N=354,354,359,228,110: number analyzed (Participants) | 354 | 354 | 359 | 228 | 110
  1M aft Inj4:PMB2948[B24]1:16;N=354,354,359,228,110 | 82.8 | 83.6 | 73.8 | 32.9 | 64.5
  1M aft Inj4:PMB2948[B24]1:32;N=354,354,359,228,110: number analyzed (Participants) | 354 | 354 | 359 | 228 | 110
  1M aft Inj4:PMB2948[B24]1:32;N=354,354,359,228,110 | 60.7 | 56.2 | 47.1 | 18.0 | 33.6
  1M aft Inj4:PMB2948[B24]1:64;N=354,354,359,228,110: number analyzed (Participants) | 354 | 354 | 359 | 228 | 110
  1M aft Inj4:PMB2948[B24]1:64;N=354,354,359,228,110 | 33.3 | 26.6 | 22.6 | 10.5 | 12.7
  1M aft Inj4:PMB2948 1:128;N=354,354,359,228,110: number analyzed (Participants) | 354 | 354 | 359 | 228 | 110
  1M aft Inj4:PMB2948 1:128;N=354,354,359,228,110 | 13.0 | 10.5 | 7.2 | 3.1 | 6.4
  Before Inj1:PMB2707[B44]1:4;N=363,357,370,241,113: number analyzed (Participants) | 363 | 357 | 370 | 241 | 113
  Before Inj1:PMB2707[B44]1:4;N=363,357,370,241,113 | 7.7 | 7.8 | 7.8 | 8.3 | 7.1
  Before Inj1:PMB2707[B44]1:16;N=363,357,370,241,113: number analyzed (Participants) | 363 | 357 | 370 | 241 | 113
  Before Inj1:PMB2707[B44]1:16;N=363,357,370,241,113 | 3.6 | 5.0 | 4.9 | 6.6 | 4.4
  Before Inj1:PMB2707[B44]1:32;N=363,357,370,241,113: number analyzed (Participants) | 363 | 357 | 370 | 241 | 113
  Before Inj1:PMB2707[B44]1:32;N=363,357,370,241,113 | 3.0 | 2.5 | 3.5 | 2.9 | 3.5
  Before Inj1:PMB2707[B44]1:64;N=363,357,370,241,113: number analyzed (Participants) | 363 | 357 | 370 | 241 | 113
  Before Inj1:PMB2707[B44]1:64;N=363,357,370,241,113 | 0.6 | 1.4 | 1.4 | 1.2 | 0.9
  Before Inj1:PMB2707 1:128;N=363,357,370,241,113: number analyzed (Participants) | 363 | 357 | 370 | 241 | 113
  Before Inj1:PMB2707 1:128;N=363,357,370,241,113 | 0.0 | 0.3 | 0.3 | 0.8 | 0.0
  1M aft Inj2:PMB2707[B44]1:4;N=341,345,349,225,111: number analyzed (Participants) | 341 | 345 | 349 | 225 | 111
  1M aft Inj2:PMB2707[B44]1:4;N=341,345,349,225,111 | 57.5 | 17.7 | 20.6 | 20.4 | 5.4
  1M aft Inj2:PMB2707[B44]1:16;N=341,345,349,225,111: number analyzed (Participants) | 341 | 345 | 349 | 225 | 111
  1M aft Inj2:PMB2707[B44]1:16;N=341,345,349,225,111 | 47.2 | 13.6 | 14.0 | 14.2 | 4.5
  1M aft Inj2:PMB2707[B44]1:32;N=341,345,349,225,111: number analyzed (Participants) | 341 | 345 | 349 | 225 | 111
  1M aft Inj2:PMB2707[B44]1:32;N=341,345,349,225,111 | 32.0 | 9.9 | 8.3 | 9.8 | 3.6
  1M aft Inj2:PMB2707[B44]1:64;N=341,345,349,225,111: number analyzed (Participants) | 341 | 345 | 349 | 225 | 111
  1M aft Inj2:PMB2707[B44]1:64;N=341,345,349,225,111 | 18.8 | 4.1 | 5.2 | 6.2 | 0.9
  1M aft Inj2:PMB2707 1:128;N=341,345,349,225,111: number analyzed (Participants) | 341 | 345 | 349 | 225 | 111
  1M aft Inj2:PMB2707 1:128;N=341,345,349,225,111 | 10.0 | 1.7 | 3.7 | 4.0 | 0.0
  1M aft Inj3:PMB2707[B44]1:4;N=333,331,341,234,105: number analyzed (Participants) | 333 | 331 | 341 | 234 | 105
  1M aft Inj3:PMB2707[B44]1:4;N=333,331,341,234,105 | 39.0 | 65.9 | 15.5 | 73.5 | 28.6
  1M aft Inj3:PMB2707[B44]1:16;N=333,331,341,234,105: number analyzed (Participants) | 333 | 331 | 341 | 234 | 105
  1M aft Inj3:PMB2707[B44]1:16;N=333,331,341,234,105 | 30.3 | 58.6 | 10.9 | 64.5 | 21.0
  1M aft Inj3:PMB2707[B44]1:32;N=333,331,341,234,105: number analyzed (Participants) | 333 | 331 | 341 | 234 | 105
  1M aft Inj3:PMB2707[B44]1:32;N=333,331,341,234,105 | 18.6 | 39.0 | 5.9 | 42.3 | 13.3
  1M aft Inj3:PMB2707[B44]1:64;N=333,331,341,234,105: number analyzed (Participants) | 333 | 331 | 341 | 234 | 105
  1M aft Inj3:PMB2707[B44]1:64;N=333,331,341,234,105 | 11.4 | 22.7 | 3.8 | 24.4 | 7.6
  1M aft Inj3:PMB2707 1:128;N=333,331,341,234,105: number analyzed (Participants) | 333 | 331 | 341 | 234 | 105
  1M aft Inj3:PMB2707 1:128;N=333,331,341,234,105 | 6.3 | 7.9 | 2.6 | 14.1 | 3.8
  1M aft Inj4:PMB2707[B44]1:4;N=356,352,356,230,111: number analyzed (Participants) | 356 | 352 | 356 | 230 | 111
  1M aft Inj4:PMB2707[B44]1:4;N=356,352,356,230,111 | 89.3 | 87.8 | 78.9 | 26.1 | 73.0
  1M aft Inj4:PMB2707[B44]1:16;N=356,352,356,230,111: number analyzed (Participants) | 356 | 352 | 356 | 230 | 111
  1M aft Inj4:PMB2707[B44]1:16;N=356,352,356,230,111 | 84.8 | 83.8 | 70.8 | 19.1 | 66.7
  1M aft Inj4:PMB2707[B44]1:32;N=356,352,356,230,111: number analyzed (Participants) | 356 | 352 | 356 | 230 | 111
  1M aft Inj4:PMB2707[B44]1:32;N=356,352,356,230,111 | 68.5 | 65.3 | 49.2 | 10.0 | 39.6
  1M aft Inj4:PMB2707[B44]1:64;N=356,352,356,230,111: number analyzed (Participants) | 356 | 352 | 356 | 230 | 111
  1M aft Inj4:PMB2707[B44]1:64;N=356,352,356,230,111 | 46.6 | 42.3 | 27.8 | 5.2 | 20.7
  1M aft Inj4:PMB2707 1:128;N=356,352,356,230,111: number analyzed (Participants) | 356 | 352 | 356 | 230 | 111
  1M aft Inj4:PMB2707 1:128;N=356,352,356,230,111 | 27.5 | 22.7 | 13.8 | 3.9 | 9.0

7. Other Pre Specified Outcome: Percentage of Participants Achieving At Least 4-fold Increase in hSBA Titer
Time Frame: 1 month after Injection 2, 3, 4
Population: Results were not reported because a decision was made a priori that, although the fold rise outcome measure will still be performed, it will not be performed as a secondary outcome measure. Therefore it was moved from a secondary outcome measure in an earlier protocol version to an exploratory outcome measure in the final protocol.
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE reported from Injection 1 to 1 month after last administration of investigational product (bivalent rLP2086/saline). SAE reported from Injection 1 to 6 months after last of investigational product (bivalent rLP2086/saline)
Description: Some participants randomized to receive vaccination as per Groups 1, 2 or 4 schedules actually received vaccination as per Group 3 schedule. One participant was not randomized but received Saline at Injection 1 and was included in Group 5. Participants have been presented as per actual administration schedule received.
Arm/Group | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month)
Serious Adverse Events (participants affected / at risk) | 12/426 | 14/414 | 7/451 | 7/277 | 3/144
Other Adverse Events (participants affected / at risk) | 113/426 | 115/414 | 114/451 | 72/277 | 43/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) (N=426) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) (N=414) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) (N=451) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) (N=277) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month) (N=144)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1:rLP2086(0-,1-,6- Month)+Saline(2- Month) (N=426) | Group 2:rLP2086(0-,2-,6- Month)+Saline(1- Month) (N=414) | Group 3: rLP2086(0-,6- Month)+Saline(1-,2- Month) (N=451) | Group 4: rLP2086(0-,2- Month)+Saline(1-,6- Month) (N=277) | Group 5: rLP2086(2-,6- Month)+ Saline(0-,1- Month) (N=144)
Injection site pain (General disorders) | 6 | 4 | 3 | 6 | 1
Pyrexia (General disorders) | 7 | 3 | 4 | 3 | 3
Fatigue (General disorders) | 5 | 5 | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 43 | 32 | 25 | 21 | 8
Pharyngitis (Infections and infestations) | 20 | 21 | 20 | 14 | 7
Upper respiratory tract infection (Infections and infestations) | 9 | 14 | 12 | 6 | 3
Gastroenteritis (Infections and infestations) | 10 | 10 | 14 | 6 | 3
Tonsillitis (Infections and infestations) | 10 | 11 | 9 | 8 | 2
Sinusitis (Infections and infestations) | 7 | 6 | 7 | 2 | 3
Bronchitis (Infections and infestations) | 4 | 5 | 9 | 0 | 2
Urinary tract infection (Infections and infestations) | 5 | 4 | 4 | 2 | 1
Rhinitis (Infections and infestations) | 3 | 4 | 3 | 3 | 2
Otitis media (Infections and infestations) | 0 | 3 | 4 | 0 | 2
Acute tonsillitis (Infections and infestations) | 0 | 4 | 1 | 3 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 5 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 10 | 3 | 5 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 4 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 2 | 1 | 2
Headache (Nervous system disorders) | 13 | 12 | 11 | 6 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.